CLINICAL TRIAL: NCT04073277
Title: Study on Improving Acupuncture Needles and Physical Properties of Acupoints With Supercritical Fluid
Brief Title: Acupuncture Needle Modified With Supercritical Fluid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMRPG8G0331
Record Dates: First submitted 2019-08-26; First posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2018-07

CONDITIONS: Healthy Participants
Keywords: Acupuncture needle; Supercritical fluid; De-qi; Chinese medicine

STUDY DESIGN:
Intervention Model Description: This was a double-blinded prospective cohort study. The acupuncture needles were first separated into two groups. One group of needles was subjected to SCF-N treatment while the other was not. The needles were then randomly analyzed with scanning electron microscope and energy dispersive X-ray spectroscopy to ensure quality and minimize experimental error. For each participant, one hand was randomly assigned to the treatment group with SCF-N-treated acupuncture needles and the other hand was assigned to the control group with the stainless steel needles. The time interval between the acupuncture treatment of the two groups was about two hours. In order to examine and distinguish the difference between the two groups, de-qi VAS score was recorded by the volunteers during needle insertion and the electrical resistance by electrical measurement.
Who Masked: Participant, Outcomes Assessor
Masking Description: The gross appearance of the two groups of needles were the same. They could be identified under microscope only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCF-N-treated needle acupuncture (Experimental): For each participant, one hand was randomly assigned to the experimental group with SCF-N-treated needle acupuncture .
  Interventions: Device: SCF-N-treated needles
- untreated needle acupuncture (Sham Comparator): The other hand of participant in experimental group was assigned to the control group with untreated needle acupuncture.
  Interventions: Device: Untreated needles

INTERVENTIONS:
Device: SCF-N-treated needles — The SCF-N-treated needles were used for acupuncture at LI 4 (Hegu) and LI 11 (Quchi) acupoints in the experimental groups..
  Arms: SCF-N-treated needle acupuncture
Device: Untreated needles — he untreated needles were used for acupuncture at LI 4 (Hegu) and LI 11 (Quchi) acupoints in the control groups.
  Arms: untreated needle acupuncture

SUMMARY:
Objective: To compare the differences in the needling sensation with acupuncture needles surface treated with nitrogen applied supercritical fluid (SCF-N) and stainless steel needles.

Materials and Methods: This was a double-blind prospective cohort study. The acupuncture needles were randomly used in this experiment, including the SCF-N-treated needles and the control stainless steel needles. LI 4 (Hegu) and LI 11 (Quchi) acupuncture points in the Yangming Large Intestine Meridian of Hand were treated. Physical electrical resistance , scanning electron microscopy, energy dispersive spectrometry, and visual analog scale score including the sensations of soreness, numbness, distention, and heaviness were assessed.

DETAILED DESCRIPTION:
This was a double-blinded prospective cohort study. The acupuncture needles were first separated into two groups. One group of needles was subjected to SCF-N treatment while the other was not. The needles were then randomly analyzed with scanning electron microscope and energy dispersive X-ray spectroscopy to ensure quality and minimize experimental error. For each participant, one hand was randomly assigned to the treatment group with SCF-N-treated acupuncture needles and the other hand was assigned to the control group with the stainless steel needles. The time interval between the acupuncture treatment of the two groups was about two hours. In order to examine and distinguish the difference between the two groups, de-qi VAS score was recorded by the volunteers during needle insertion and the electrical resistance by electrical measurement.

The acupuncture needles used in this experiment, including the SCF-N-treated needles and the control stainless steel needles, were produced under the same conditions, in the same factory (Dong Bang acupuncture Inc.), and on the same day, to minimize experimental error.

The process of SCF treatment:. First, the stainless steel chamber and quartz carrier were sterilized using alcohol and autoclaving. Next, the needles were placed on the quartz carrier with the tip pointing upwards and then placed in the chamber and covered. Carbon dioxide was used to remove atmospheric components from the chamber and required volume of ammonia gas was passed. The pressure was increased up to 3000 pound per square inch(psi) and temperature up to 120℃. An hour later, the pressure was relieved and the process of SCF treatment completed. After completion of the treatment, the needles were then randomly selected for material analysis and electrical measurement. Following this, the needles were stored in a vacuum bag. This was done to reduce the influence of atmospheric contaminants on the needles after treatment, resulting in oxidation and rusting. Finally, there would be heterogeneous contact between the inorganic metal and the acupuncture needle. Hence, nitrogen was selected as the main agent for SCF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer aged 20 to 40 years
* Provided informed consent

Exclusion Criteria:

* Women with pregnancy or breast feeding
* Bleeding tendencies (platelet counts less than 20000 and/or thrombocytopenic purpura)
* Volunteers with chronic medical conditions and anti-coagulants use
* Volunteers with pacemakers
* Fasting
* Unwilling to provide informed consent

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Resistance of the meridian | immediately after acupuncture needling
  Electrical resistance was measured by applying a fixed electric current (110 µA) for 1 second and recording the I-V curve. A linear relationship of voltage=current x resistance was expected. The analyzer used in this experiment was Agilent B1500, a semi-conductor analyzer able to measure electrical resistance with high accuracy.

SECONDARY OUTCOMES:
Modified Visual Analog Scale (VAS) Score | immediately after acupuncture needling
  The VAS score was used to assess the needling sensations of de-qi, i.e. distension, soreness, heaviness, or numbness. VAS score 0 indicated no sensation, while VAS 10 indicated the strongest sensation.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan